CLINICAL TRIAL: NCT05165901
Title: Clinical Effect of LG Medipain for Managing Chronic Pain Disorders: A Prospective Observational Study
Brief Title: Clinical Effect of LG Medipain for Managing Chronic Pain Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeeyoun Moon (Other)
Responsible Party: Sponsor-Investigator, Jeeyoun Moon, Chief director, pain management center, Seoul National University Hospital, Seoul National University
Organization: Seoul National University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2110-017-1260
Record Dates: First submitted 2021-11-01; First posted 2021-12-21 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Neuropathic Pain; Pain; Refractory Pain; Chronic Pain
MeSH Terms: conditions — Neuralgia; Pain; Pain, Intractable; Chronic Pain

STUDY DESIGN:
Intervention Model Description: 3 different chronic pain classification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nociceptive pain (Experimental): patients with joint pain (knee and shoulder), myofascial pain syndrome
  Interventions: Device: Scrambler Therapy
- Neuropathic pain (Experimental): patients with postherpetic neuralgia, peripheral nerve injury (CRPS type II, brachial plexopathy, nerve entrapment syndrome)
  Interventions: Device: Scrambler Therapy
- Mixed pain (Experimental): patients with spine or SIJ origin back and buttock pain or neck pain and SPINE-origin back pain과 neck pain, SIJ-origin back and buttock pain
  Interventions: Device: Scrambler Therapy

INTERVENTIONS:
Device: Scrambler Therapy — LG Medipain is a type of non-invasive neuromodulation.

SUMMARY:
Scrambler Therapy is a type of non-invasive neuromodulation. According to the researches that studied the effects of the existing Scrambler therapy, 10 times of Scrambler Therapy showed a significant pain relief lasting for more than 1-3 months in various pain disorders such as post-herpetic neuralgia, cancer-related neuropathic pain, and mixed pain. No treatment-related side effects have been reported in Scrambler therapy conducted in previous studies.

The most inconvenient thing about Scrambler Therapy is that it has to be treated more than 10 times during specific period, so frequent visits to the hospital for treatment linked to the higher burden for the patient's cost and even those are not fully covered by the government's insurance. To reduce this discomfort and expand the range of treatment in the era of Corona of untact treatment, LG Electronics devised a home self-scrambler treatment device for pain patients.

The LG Medipain device has the same treatment function as the existing hospital Scrambler treatment device, but there has been no study on its efficacy and safety. Therefore, the investigators want to conduct this research and find out about the safety and equal efficiency of the LG Medipain Therapy.

In this study, it is expected that pain relief and improvement of quality of life can be obtained for patients with various types of chronic pain through self-application of LG Medipain device.

DETAILED DESCRIPTION:
Scrambler Therapy is a type of non-invasive neuromodulation. Scrambler Therapy is a different type of pain treatment from the theory that converts pain signals into general sensory information (non-pain signals) generated in the human body through artificial neurons and transmits them to the CNS through A-delta and C-nerve fibers, which are pain-transmitting nerve fibers. The non-pain signal converted through Scrambler Therapy exhibits a pain modulatory effect through CNS education, and eventually, the pain signal is continuously disturbed into a pain-free signal, resulting in pain relief. This will function to normalize neuronal plasticity, the cause of chronic pain, which is different from existing pain treatments based on the gate control theory that temporarily blocks or alleviates the recognition of pain stimuli in the CNS.

Scrambler therapy is similar to the existing TENS treatment, but the treatment process is very different from TENS. TENS is a principle that replaces the delivery of pain stimulus to the brain with a stimulus other than pain stimulus and transmits it to the brain. However, Scrambler Therapy is a treatment that reduces the perception of pain in the brain by scrambling the conversion of pain stimulation into electrical signals in the peripheral nerves, similar to TENS, but can convert pain signals into pain-free signals through repetitive brain learning. So to speak, the investigators could state that it is a treatment method that fundamentally suppresses the generation of pain signals.

According to the researches that studied the effects of the existing Scrambler therapy, 10 times of Scrambler Therapy showed a significant pain relief lasting for more than 1-3 months in various pain disorders such as post-herpetic neuralgia, cancer-related neuropathic pain, and mixed pain. No treatment-related side effects have been reported in Scrambler therapy conducted in previous studies.

The most inconvenient thing about Scrambler Therapy is that it has to be treated more than 10 times during specific period, so frequent visits to the hospital for treatment linked to the higher burden for the patient's cost and even those are not fully covered by the government's insurance. To reduce this discomfort and expand the range of treatment in the era of Corona of untact treatment, LG Electronics devised a home self-scrambler treatment device, LG Medipain for pain patients.

While the hospital Scrambler Therapy device uses up to 5 channels (with 10 patches attached) for treatment and the size of the machine is large, the LG Medipain device uses 2 channels (up to 4 patches attached) and is portable and easy to use which is designed to be convenient. The LG Medipain device has the same treatment function as the existing hospital Scrambler treatment device, but there has been no study on its efficacy and safety. Therefore, the investigators want to conduct this research and find out about the safety and equal efficiency of the LG Medipain Therapy. In addition, in order to explore the mechanism of LG Medipain treatment, 30 patients who responded to treatment will be selected and the investigators have plan to examine their EEG waveform of 32 channel with their consents.

After 2 weeks of applying the LG Medipain Therapy for various chronic pain diseases, meaningful (MCD 30% for each group) pain relief effect will be obtained. The purpose of this study is to check whether pain relief can be obtained after 2 weeks of applying 10 times of the LG Medipain therapy for various chronic pain diseases. The secondary purpose of this study is to compare the pain and related-function improvement effects of the LG Medipain Therapy by pain classification. Scrambler treatment has been reported to have a pain relief effect on postherpetic neuralgia, various cancer pains, and musculoskeletal pain through basic 10 applications. In this study, it is expected that pain relief and improvement of quality of life can be obtained for patients with various types of chronic pain through self-application of the LG Medipain device.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain disease (pain over 3 months) as an adult 19 years of age or older
* Patients with 11-pointed NRS pain score ≥ 4 for the corresponding pain on the day of admission
* Patients taking oral pain treatment drugs in the same type and dose up to 1 month before participating in the study, and taking the same medication until 1 month after participating in the study (at the time of obtaining the primary endpoint)
* Those who voluntarily and in writing consent to participate in the study
* A person who has agreed in writing to return the Scrambler Therapy device
* By the classification of pain disorder, patients include with nociceptive pain such as joint pain, myofascial pain syndrome and with neuropathic pain such as postherpetic neuralgia, peripheral nerve injury and nerve entrapment syndrome and with mixed pain.

Exclusion Criteria:

* Refusal of the patient
* In case pain relief effect was not obtained in the past Scrambler Therapy
* Patients currently undergoing Scrambler therapy for pain control at outpatient clinics at the Pain Center
* Patients who had previously taken Scrambler Therapy 6 months before participating in the study
* In case of systemic infection or local infection in the area around the treatment (the patch attachment site)
* Patients who has cognitive decline that cannot understand the contents of the Numeric Pain Rating (NRS), questionnaire, and scrambler self application method
* If it is difficult to self-administer 10 scrambler treatments for 2 weeks during the treatment period
* Women during pregnancy
* In case of implantation of a pacemaker, brain stimulator, etc.
* Those who are not suitable for this clinical trial under the judgment of other investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain relief scoreobtained after 2 weeks of applying | after 2 weeks of applying
  Pain relief by NRS(Numeric rating scale): from 0(no pain) to 10(worst pain possible)

SECONDARY OUTCOMES:
The painDETECT questionnaire (PD-Q) | during 1 year of treatment
  The painDETECT questionnaire (PD-Q) for neuropathic pain score assessment
EuroQol-5 dimention(EQ-5D) | during 1 year of treatment
  EuroQol-5 dimention(EQ-5D) for describing and valuing the health of life
patient global impression of change (PGIC) | during 1 year of treatment
  patient global impression of change (PGIC) in self-report 5 scale reflects a patient's belief about the efficacy of treatment
Insomnia Severity Index | during 1 year of treatment
  Insomnia Severity Index for assessing sleep difficulty
Oswestry Disability Index(ODI) | during 1 year of treatment
  Oswestry Disability Index(ODI) for back & neck functional disability
The Western Ontario and McMaster Universities(WOMAC) Index | during 1 year of treatment
  The Western Ontario and McMaster Universities(WOMAC) Index to evaluate the patient's Hip and Knee Osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Yoon Moon, Pf, Study Director — Seoul national universitiy Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No